CLINICAL TRIAL: NCT02003170
Title: Etiology and Early Diagnosis of Neurodevelopmental Disorders
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 136272
Record Dates: First submitted 2013-11-25; First posted 2013-12-06 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Neurodevelopmental Disorders
Keywords: Autism; Autism Spectrum Disorder (ASD); Pervasive Developmental Disorder (PDD); Developmental delays; Genetic disorder; Mitochondrial disorder
MeSH Terms: conditions — Neurodevelopmental Disorders; Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Genetic Diseases, Inborn; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, cerebrospinal fluid, muscle, and skin samples may be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurodevelopmental Disorders: Children who present to various Arkansas Children's Hospital clinics for standard care related to neurodevelopmental disorders.

SUMMARY:
The purpose of this study is to systematically evaluate the results of medical investigations to identify symptom and biological patterns and common etiologies of neurodevelopmental disorders.

DETAILED DESCRIPTION:
Although neurodevelopmental disorders are very prevalent (for example Autism affects 1 out of every 88 children and dyslexia affects up to 15% of the population), the etiology of such disorders is not known. The purpose of this investigation is to identify common etiologies of neurodevelopmental disorders (i.e., speech delay, global developmental delay, autism) and determine if it is possible to find early indicators of the diagnosis and foster the potential for a better prognosis of these disorders. At this time the investigators examine patients with neurodevelopment disorders with various medical investigations, but the results of these investigations are not systematically evaluated. One of the goals of this research is to systematically examine this information in order to identify patterns of test abnormalities that have not been previously described. Another goal of this research is to identify the common etiologies typically identified by the medical evaluation, so we can further refine our approach. In addition, the investigators now have the ability to evaluate biological samples for biomarkers that have potential to be diagnostically useful.

ELIGIBILITY:
Inclusion Criteria:

* Neurodevelopmental delays
* Clinical visit at an Arkansas Children's Hospital Outpatient clinic

Exclusion Criteria:

* none

Ages: 0 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children who present to various Arkansas Children's Hospital Outpatient clinics for standard care related to neurodevelopmental disorders.
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2012-05; Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Medical abnormalities associated with specific neurodevelopmental disorders | up to 7 years
  It is unknown if a specific set of biological abnormalities contribute to the formation of many types of neurodevelopmental disorders. The study is intended to identify the relationship between biological abnormalities and neurodevelopmental disorders

SECONDARY OUTCOMES:
Biomarkers associated with neurodevelopmental disorders | up to 7 years
  It is unknown if a specific biomarkers are associated with specific neurodevelopmental disorders. The study is intended to identify the relationship between biological abnormalities and neurodevelopmental disorders
Treatments associated with neurodevelopmental disorders | up to 7 years
  Various behavioral and medical treatments are used for many types of neurodevelopmental disorders but the effectiveness for many of these treatments is not known. The study is intended to identify the relationship between biological abnormalities (and their treatments) and neurodevelopmental disorders

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Rose, PhD., Principal Investigator — Arkansas Children's Hospital Research Instisute; UAMS
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Frye RE, Lionnard L, Singh I, Karim MA, Chajra H, Frechet M, Kissa K, Racine V, Ammanamanchi A, McCarty PJ, Delhey L, Tippett M, Rose S, Aouacheria A. Mitochondrial morphology is associated with respiratory chain uncoupling in autism spectrum disorder. Transl Psychiatry. 2021 Oct 13;11(1):527. doi: 10.1038/s41398-021-01647-6. PMID 34645790
- See also: To see a list of current clinical Trials at Arkansas Children's Hospital, click here!! — https://www.archildrens.org/programs-services/clinical-trials/enrolling-studies